CLINICAL TRIAL: NCT02023346
Title: Prognostic Awareness and Patient-Physician Communication in Malignant Glioma
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 13-253
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Malignant Glioma
Keywords: Patient-Physician Communication; Brain cancer; 13-253
MeSH Terms: conditions — Glioma; Brain Neoplasms | interventions — Surveys and Questionnaires; Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Malignant Glioma patients: This is a cross-sectional study of patients with MG who are admitted to the inpatient Neurology service at MSKCC. We anticipate that participants will be accrued over approximately 18-24 months. All patients with MG admitted to Neurology, will be screened for eligibility and willingness to participate in the study.
  Interventions: Behavioral: surveys and cognitive tests

INTERVENTIONS:
Behavioral: surveys and cognitive tests

SUMMARY:
The purpose of this study is to learn more about the understanding patients with brain tumors have of their disease and their communication with their physician. Ultimately, we hope to use these findings to improve communication between patients and their doctors.

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion Criteria

* Age greater than or equal to 18
* Diagnosis of any WHO grade III or IV glioma
* Admitted to the inpatient Neurology service
* Has had at least one outpatient visit with a neuro-oncologist at MSKCC Fluent in English

Caregiver Inclusion Criteria

* Age greater than or equal to 18
* Identified by the patient as a relative, friend, or partner with whom he or she has a significant relationship and who provides him or her physical or emotional assistance.
* The patient has himself or herself agreed to participate in this study

Exclusion Criteria:

Patient Exclusion Criteria

* A patient will be excluded if the Glasgow Coma Scale is less than 15. The patient must be oriented to self, age, place, and year, and month.
* Aphasia precluding comprehension and verbalization of consent to participate
* Patients who cannot verbally demonstrate their understanding of the risks, benefits, and alternatives to participating in the study. This evaluation will take place for otherwise eligible and willing participants, and it will be performed by the NP or MD clinician who is obtaining informed consent and will be documented in the medical record.

Caregiver Exclusion Criteria

* No eligible caregivers who can complete the brief assessment in person or via telephone will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the inpatient Neurology service. Caregivers will be recruited from either the inpatient Neurology service (if they are physically present at the hospital at the time of the patient's consent to participate) or via telephone communication (if not physically present at the time of patient consent).
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
measure prognostic awareness | 2 years
  Prognostic awareness (PA) will be measured using the Chochinov Prognostic Awareness Scale. This scale classifies patients into three categories of awareness: full, limited, or no awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Eli Diamond, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memoral Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/